CLINICAL TRIAL: NCT02125526
Title: Survival Improvement in Extensive Myocardial Infarction With PERsistent Ischemia Following Intra-aortic Balloon Pump Implantation
Brief Title: Intra-aortic Balloon Pump in Extensive Myocardial Infarction With Persistent Ischemia
Acronym: SEMPER FI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokien van Nunen (Other)
Collaborators: Stichting Toegepaste Wetenschappen (project number 11052) (Unknown); Maquet Cardiovascular (Industry)
Responsible Party: Sponsor-Investigator, Lokien van Nunen, MD, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IABPinPI; STW-11052 (Other: Stichting Toegepaste Wetenschappen)
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Acute Myocardial Infarction; Persisting Ischemia; No Reflow
Keywords: Acute myocardial infarction; Persisting ischemia; No reflow; Intra-aortic balloon pump; Exhausted autoregulation
MeSH Terms: interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IABP group (Active Comparator): After primary percutaneous coronary intervention, IABP will be implanted for 12-24 hours to alleviate persisting ischemia
  Interventions: Device: Intra-aortic balloon pump
- Control group (No Intervention): After primary percutaneous coronary intervention, this group undergoes standard treatment according to the guidelines

INTERVENTIONS:
Device: Intra-aortic balloon pump — The intra-aortic balloon pump is placed in the descending thoracic aorta and inflates and deflates in synchrony with the cardiac cycle, providing diastolic augmentation and improving coronary blood flow, while deflating before systole, providing afterload and workload reduction for the myocardium.
  Other Names: IABP; Intra-aortic balloon counterpulsation
  Arms: IABP group

SUMMARY:
Patients presenting with large myocardial infarction and signs of persistent ischemia after successful percutaneous coronary intervention, have a poor prognosis with respect to outcome and development of heart failure in the future.

The hypothesis of this study is that in patients in whom persistent ischemia is present, use of intra-aortic balloon pump will be beneficial and improve outcome.

DETAILED DESCRIPTION:
In some patients presenting with large myocardial infarction and poor hemodynamic condition, intra-aortic balloon counterpulsation is effective in alleviating cardiogenic shock. In others, the use of intra-aortic balloon pump has no effect at all. The investigators believe this is dependent on the presence of persisting ischemia after successful epicardial reperfusion, known as no-reflow.

In the presence of persisting ischemia, the investigators believe us of the intra-aortic balloon pump will relieve ischemia and improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* Acute ST-segment elevation myocardial infarction with summed ST-segment deviation ≥15 mm.
* Insufficient ST-segment resolution (<50%) on the ECG made 10-30 minutes after the primary PCI in the catheterization laboratory.

Exclusion Criteria:

* Initial summed ST-segment deviation less than 15 mm
* ST-segment resolution > 50% on the ECG performed in the catheterization laboratory
* Chest pain onset less than 2 or more than 8 hours before arrival
* Severe aortic valve stenosis/regurgitation
* Aortic abnormalities prohibitive for use of intra aortic balloon pump
* Full blown cardiogenic shock with immediate requirement of left ventricular assist device as judged necessary by the operator
* Inability to provide informed consent
* Pregnancy
* Inability to perform coronary angiography by the femoral approach

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of mortality, necessity for mechanical support due to hemodynamic deterioration, and hospital admission for heart failure | 6 months
All-cause mortality | 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nico H.J. Pijls, MD PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Lokien X van Nunen, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] van Nunen LX, van 't Veer M, Schampaert S, Steerneman BJ, Rutten MC, van de Vosse FN, Pijls NH. Intra-aortic balloon counterpulsation in acute myocardial infarction: old and emerging indications. Neth Heart J. 2013 Dec;21(12):554-60. doi: 10.1007/s12471-013-0485-9. PMID 24170231